CLINICAL TRIAL: NCT00635661
Title: A Comparison of the Stroke Rehabilitation Assessment of Movement, the Functional Independence Measure and the Stroke Impact Scale
Brief Title: Assessment of the Stroke Rehabilitation Assessment of Movement as a Clinical Tool
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: NYU Langone Health (Other)
Responsible Party: Principal Investigator, Gary Brooks, Associate Professor, State University of New York - Upstate Medical University
Other Study IDs: IRBPHS-5535
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Results first posted 2012-03-02 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-01

CONDITIONS: Stroke
Keywords: function; disability
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Stroke Rehabilitation Assessment of Movement (STREAM) is a relatively new measurement tool, which measures specific movement deficits (impairments) caused by a stroke. The STREAM is used to evaluate recovery of voluntary movement and basic mobility following the onset of a stroke. Several important clinical measurement properties of the STREAM remain to be explored, including its ability to measure impairments and clinical change in acute rehabilitation patients in the USA. We hypothesize that the STREAM will be able to detect and quantify a statistically significant change in the motor abilities of stroke patients from admission to discharge. An additional aim of the study is to compare the STREAM with two accepted and widely used clinical measures of function and disability, the Stroke Impact Scale (SIS)and the Functional Independence Measure (FIM). By linking movement deficits that are commonly assessed by physical therapists with measures of function and disability, the impact of the movement deficits can be understood.

ELIGIBILITY:
Inclusion Criteria:

* comprehension of English
* age 18 and older
* first-time stroke
* receiving in-patient rehabilitation at the Rusk Institute of Rehabilitation Medicine, New York, NY

Exclusion Criteria:

* hemorrhagic stroke
* brain stem or cerebellar infarct
* other pre-existing neurologic conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who have sustained an ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Ward, DPT, Principal Investigator — NYU Medical Center, Rusk Institute
Locations (1):
- Rusk Institute of Rehabilitation Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Participants: The study participants comprise the cohort on whom data are collected. All participants received usual rehabilitation care following admission. No experimental intervention(s) were provided.
Period: Overall Study
Arm/Group | Study Participants
Started | 34
Completed | 30
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Study Participants
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 66.1 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Stroke Rehabilitation Assessment of Movement (STREAM)
Description: The STREAM measures quality of movements in the arm and leg, and the quality of mobility during important functional tasks, such as walking 10 feet. There are 10 items for each of the 3 assessments (arm, leg and mobility), resulting in a total of 30 items. Each item is rated on a scale of 0 = unable to perform, to 2 or 3 = normal movement. Ratings on the 30 items are added together for a total score which is divided by the total number of items resulting in a percentage score: minimum=0, maximum=100, range=100 The score reported is mean +/- standard deviation of discharge STREAM scores.
Time Frame: 4 weeks
Population: 34 participants were enrolled, 4 participants were dropped from the study resulting in 30 participants providing data for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Participants
Number analyzed (Participants) | 30
units on a scale | 73.1 (26.1)

ADVERSE EVENTS:
Arm/Group | Study Participants
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No